CLINICAL TRIAL: NCT00714298
Title: Analyse en médecine d'Urgence d'Une stratégie d'Utilisation combinée de Deux Marqueurs Biologiques Dans le Diagnostic de Syndrome Coronaire Aigu Non ST+: étude Des Performances de la Heart-Fatty Acid Binding Protein et de l' Ischemia Modified Albumin dès la première Heure de Prise en Charge
Brief Title: Diagnostic Value of Heart-Fatty Acid Binding Protein and Ischemia Modified Albumin as Biochemical Markers on Non ST Segment Elevation Acute Coronary Syndrome at the Emergency Room.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Nathalie ROQUES, U H TOULOUSE
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0503408; PHRC
Record Dates: First submitted 2008-07-07; First posted 2008-07-14 (Estimated); Last update posted 2008-07-14 (Estimated); Status verified 2008-07

CONDITIONS: Acute Coronary Syndrome
Keywords: biological markers; emergency service hospital; heart fatty acid binding protein; ischemia modified albumin
MeSH Terms: conditions — Acute Coronary Syndrome; Emergencies | interventions — ischemia-modified albumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Initial heart fatty acid binding protein and ischemia modified albumin will be measured after patient's arrival in the emergency room. Treating physicians, biologist physician will be blinded to the results of the markers.
  Interventions: Other: Measure of Initial heart fatty acid binding protein and ischemia modified albumin

INTERVENTIONS:
Other: Measure of Initial heart fatty acid binding protein and ischemia modified albumin — Initial heart fatty acid binding protein and ischemia modified albumin will be measured after patient's arrival in the emergency room. The aim of the study is to analyse the predictive value of association of heart fatty binding protein and ischemia modified albumin for non ST segment elevation acute coronary syndrome diagnosis in the first hour of management in the emergency room.Treating physicians, biologist physician will be blinded to the results of the markers.

SUMMARY:
Early diagnostic of non ST elevation coronary syndrome in patients admitted to the emergency room is difficult. Two news biochemical markers have been assessed and studies have suggested that heart fatty binding protein and ischemia modified albumin are early markers of myocardial necrosis and myocardial ischemia. The aim of the study is to analyse the predictive value of association of heart fatty binding protein and ischemia modified albumin for non ST segment elevation acute coronary syndrome diagnosis in the first hour of management in the emergency room.

DETAILED DESCRIPTION:
Early diagnostic of non ST elevation coronary syndrome (ACS) in patients admitted to the emergency room is difficult. Two news biochemical markers have been assessed and studies have suggested that heart fatty binding protein and ischemia modified albumin are early markers of myocardial necrosis and myocardial ischemia.

Study objective: The aim of the study is to analyse the predictive value of association of heart fatty binding protein and ischemia modified albumin for non ST segment elevation ACS diagnosis in the first hour of management in emergency room.

Methods: In a prospective double blind study, initial heart fatty binding protein and ischemia modified albumin levels will be measured in consecutive patients admitted in the emergency room with chest pain and suspected non-ST elevation ACS. Data including history, physical examination, serial 12-lead ECG and troponin-I measurement at 0 and 6 hours after admission will be collected by the treating physician blinded to the result of the markers. Based on hospital diagnosis algorithm (troponin repeated measurements, treadmill test or other ischemia detection, coronarography if necessary) and follow-up at one month, patients will be classified as having or no non-ST elevation ACS by two independent physicians blinded to the results of markers. Sensitivity, specificity, positive and negative predictive values will be determined for each marker and in combined analyses.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients admitted in the emergency room with a primary complaint of chest pain evolving within 12 hours and suspected as acute coronary syndrome

Exclusion Criteria:

* patient younger than 18 years old, having an ST elevation on a 12-lead ECG, having an evident traumatic cause of chest pain or having severe communication problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2006-05; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
non ST segment elevation ACUTE coronary syndrome diagnosis | One month

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine CHARPENTIER, MD, Principal Investigator — U H TOULOUSE
Locations (1):
- Emergency department Rangueil, Toulouse, France

REFERENCES:
- [Derived] Charpentier S, Maupas-Schwalm F, Cournot M, Elbaz M, Botella JM, Lauque D. Combination of copeptin and troponin assays to rapidly rule out non-ST elevation myocardial infarction in the emergency department. Acad Emerg Med. 2012 May;19(5):517-24. doi: 10.1111/j.1553-2712.2012.01350.x. PMID 22594355
- [Derived] Charpentier S, Cournot M, Lauque D, Girardi C, Bounes V, Elbaz M, Ducasse JL. Usefulness of initial glucose level to improve acute coronary syndrome diagnosis in the emergency department. Emerg Med J. 2011 Jul;28(7):564-8. doi: 10.1136/emj.2010.094284. Epub 2010 Jul 20. PMID 20659883
- [Derived] Charpentier S, Ducasse JL, Cournot M, Maupas-Schwalm F, Elbaz M, Baixas C, Juchet H, Lang T, Lauque D. Clinical assessment of ischemia-modified albumin and heart fatty acid-binding protein in the early diagnosis of non-ST-elevation acute coronary syndrome in the emergency department. Acad Emerg Med. 2010 Jan;17(1):27-35. doi: 10.1111/j.1553-2712.2009.00614.x. PMID 20078436